CLINICAL TRIAL: NCT04284631
Title: Prognostic Value of Her2neu and EGFR in Primary Ovarian High Grade Serous Carcinoma.
Status: Completed | Type: Observational
Sponsor: Port Said University hospital (Other)
Responsible Party: Principal Investigator, Mayada saad, Lecturer of pathology, Port Said University hospital
Other Study IDs: pathology1
Record Dates: First submitted 2020-02-22; First posted 2020-02-26 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess alterations of EGFR& Her2neu expression in primary ovarian high grade serous carcinoma and its correlation with other clinicopathological parameters

DETAILED DESCRIPTION:
Ovarian cancer (OC) is the seventh most common cancer and the fifth cause of cancer death in women worldwide. The most frequent type is surface epithelial tumors. It is frequently diagnosed at advanced stages. So, it is referred to as silent killer.

Serous carcinoma is the most common and aggressive type of epithelial ovarian cancer . Serous carcinomas are currently separated into two completely different subtypes either histologically or biologically, lowg rade and high grade, based on both degree of nuclear atypia and the number of mitoses.

Current therapy is based on few traditional prognostic factors, such as tumor stage and postoperative tumor residual mass. Identification of new molecular markers could help in significant modification of treatmant improving clinical prognosis The ErbB family of tyrosine kinase receptors (epidermal growth factor (EGF) receptors) plays a role in the tumorigenesis of several types of solid tumors. The abnormal activation of these receptors has been associated with various pathological processes especially cellular transformation .

EGFR is involved in various stages of cancer growth, such as tumor initiation, angiogenesis and metastasis. Also, it participates by various pathways as a proto-oncogene in several types of cancers such as gastrointestinal and breast ones. So, it is an attractive target for oncogenic therapy HER2 protooncogene is involved in the development of many types of human cancer and is used as therapeutic target. Although the association between HER2 expression and ovarian cancer has been widely studied, the results are still controversial Therefore, in the present study we will analyze the expression of both EGFR& Her2neu in an OC tissue microarray (TMA) by immunohistochemistry, and results were be correlated to other clinicopathological parameters and prognosis.

Aim of the study:

General aim: To assess alterations of EGFR& Her2neu expression in primary ovarian high grade serous carcinoma and its correlation with other clinicopathological parameters.

Specific objectives:

1. To measure the frequency of EGFR& Her2neu immunohistochemical expression in ovarian high grade serous carcinoma.
2. To correlate between expression of EGFR& Her2neu expression and other clinicopathological parameters of ovarian high grade serous carcinoma
3. To correlate between expression of EGFR& Her2neu expression and prognosis of ovarian high grade serous carcinoma

Materials:

This cross-sectional study will be done on 54 specimens of ovarian primary high grade serous carcinoma cases who attended to Oncology Centre, Mansoura University, Mansoura, Egypt since 2012 to the end of 5 years follow up of the last patient The cases will be chosen randomly.

Methods:

1. All clinicopathological data of these cases will be collected such as Tumor size, LN metastases (N), metastasis (M), ascites, residual tumor, peritoneal deposits, recurrence, TNM staging & (FIGO) staging system.
2. Prepare hematoxylin & eosin slides to diagnose and assess other histopathological parameters such as histological type
3. Immunohistochemistry:

Sections 4μm thickness from newly formed tissue microarray blocks will be cut on coated slides then immunohistochemical staining using antibody against EGFR& Her2neu will be done.

Statistical analysis:

SPSS software version 20 (SPSS Inc., Chicago, IL) will be used for analysis. For nominal variables, proportions and X2 tests will be applied, whereas for interval variables means, standard deviations (SD), and T test and ANOVA tests will be applied where appropriate. Kaplan-Meier method will be used for survival analysis. Chi-square test was used to estimate the relation between qualitative variables. Mann-Whitney test (non-parametric t test) was used for not normally distributed quantitative data, for comparison between two groups while, comparison between three groups was done using Kruskal-Wallis test (non-parametric ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary ovarian cancer

Exclusion Criteria:

* patients with secondary ovarian cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Patients with primary ovarian cancer
Study Population: All patients undergone exploratory laparotomy for primary ovarian cancer Sections 4μm thickness from newly formed tissue microarray blocks will be cut on coated slides then immunohistochemical staining using antibody against EGFR& Her2neu will be done.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
EGFR& Her2neu expression to the grade of ovarian serous carcinoma | 2 years
  EGFR& Her2neu expression in primary ovarian high grade serous carcinoma
EGFR& Her2neu expression in primary ovarian serous carcinoma to prognosis | 5 years
  Expression of EGFR & Her2neu in primary ovarian cancer to cancer free period